CLINICAL TRIAL: NCT02331641
Title: Multiple Minor Hepatectomies Versus Major or Extended Hepatectomies for Colorectal Liver Metastases. A Propensity Score-matched Dual-institution Analysis.
Brief Title: Multiple Minor Hepatectomies Versus Major or Extended Hepatectomies for Colorectal Liver Metastases.
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: MajorVsMinorHepatectomy
Record Dates: First submitted 2014-12-29; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Liver Metastases; Colon Cancer
Keywords: hepatectomy; hepatic resection
MeSH Terms: conditions — Colonic Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major hepatectomy (MH): Patients who underwent MH for CLM instead of multiple minor hepatectomy (MMH)
  Interventions: Procedure: Hepatectomy
- Multiple minor hepatectomy (MMH): Patients who underwent MMH for CLM instead of MH
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Removal of a part of the liver
  Other Names: Hepatic resection

SUMMARY:
The performance of multiple minor hepatectomies (MMH) instead of major hepatectomies (MH) in patients with colorectal liver metastases (CLM) is object of debate. We build a study, using the propensity score matched analysis, to compare the short- and long-term outcome of the tow groups of patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate the outcome of patients with colorectal liver metastases (CLM) undergoing multiple minor hepatectomies (MMH) instead of major hepatectomies (MH). Indeed, the performance of MMH versus MH in patients with CLM is object of debate. For this purpose, the databases at two independent institutions were retrospectively reviewed. To control for confounding variable distributions, a propensity score-matched analysis 1:1 was performed, and the nearest neighbor-matching method with caliper distance of 0.01 was used. Among 554 patients, 110 patients undergoing MMH and 110 undergoing MH were matched. They were similar in baseline characteristics, comorbidities, features of the primary tumors, and CLM. Primary outcomes were short- and long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLM

Exclusion Criteria:

* Uncertain diagnosis
* Lost at follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal liver metastases (CLM) that underwent hepatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2005-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of postoperative complications after MH or MMH, graded based on the Dindo's classification (Dindo et al. Ann Surg 2004;240:205-13) | up to 90 days after surgery

SECONDARY OUTCOMES:
Long-term outcome (overall and disease-free survival) | 10 years
  Typical follow-up after surgery (until death and evidence of recurrence)